CLINICAL TRIAL: NCT06052462
Title: Disposition of [14C]-LY3556050 Following Oral Administration in Healthy Male Participants
Brief Title: A Study of Carbon-14-Labelled [14C] LY3556050 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18347; J2P-MC-LXBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-LY3556050 (Experimental): Single dose of [¹⁴C]-LY3556050 administered orally
  Interventions: Drug: [14C]-LY3556050

INTERVENTIONS:
Drug: [14C]-LY3556050 — Administered orally

SUMMARY:
The main purpose of this study is to evaluate how much of the study drug (LY3556050), administered as a single dose that has the radioactive substance 14C incorporated into it, passes from blood into urine, feces and expired air in healthy male participants. The study will also measure how much of the study drug gets into the bloodstream, how its broken down, and how long it takes the body to get rid of it. The study will last up to approximately 58 days including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are overtly healthy as determined by medical evaluation
* Have a body mass index of 18.0 to 32.0 kilograms per meter squared (kg/m²), inclusive
* Males who agree to use highly effective or effective methods of contraception

Exclusion Criteria:

* Have known allergies to LY3556050, related compounds, or any components of the formulation of LY3556050, or history of significant atopy
* Have clinically significant abnormal BP and/or pulse rate as determined by the investigator
* Have had exposure to significant diagnostic, therapeutic, or employment-related radiation within 12 months prior to dosing

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-11-04 (Actual); Study Completion 2023-11-04 (Actual)

PRIMARY OUTCOMES:
Urinary Excretion of LY3556050 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Predose up to Day 21 post dose
  Urinary Excretion of LY3556050 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Fecal Excretion of LY3556050 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Predose up to Day 21 post dose
  Fecal Excretion of LY3556050 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Curve Concentration Versus Time Curve From Time zero to Last Time Point (AUC[0-tlast]) of LY3556050 in Plasma | Predose up to Day 21 post dose
  PK: AUC(0-tlast) of LY3556050 in Plasma
PK: AUC(0-tlast) of Total Radioactivity in Plasma and Blood | Predose up to Day 21 post dose
  PK: AUC(0-tlast) of Total Radioactivity in Plasma and Blood
PK: Area Under the Curve Concentration Versus Time Curve From zero to Infinity (AUC [0-∞]) of LY3556050 in Plasma | Predose up to Day 21 post dose
  PK: AUC (0-∞) of LY3556050 in Plasma
PK: AUC (0-∞) of Total Radioactivity in Plasma and Blood | Predose up to Day 21 post dose
  PK: AUC (0-∞) of Total Radioactivity in Plasma and Blood
PK: Maximum Concentration (Cmax) of LY3556050 in Plasma | Predose up to Day 21 post dose
  PK: Cmax of LY3556050 in Plasma
PK: Cmax of Total Radioactivity in Plasma and Blood | Predose up to Day 21 post dose
  PK: Cmax of Total Radioactivity in Plasma and Blood
Total Radioactivity Recovered in Urine, Feces, and Expired Air (if applicable) | Predose up to Day 7 post dose
  Total Radioactivity Recovered in Urine, Feces, and Expired Air (if applicable)
Total Number of Metabolites of LY3556050 | Predose up to Day 7 post dose
  Total Number of Metabolites of LY3556050

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- LabCorp CRU, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No